CLINICAL TRIAL: NCT01646229
Title: Impact of Early Per-operative Use of Polymyxin-B Hemoperfusion in Septic Patients Undergoing Emergent Abdominal Surgery
Brief Title: Impact of Early Peri-operative Use of Polymyxin-B Hemoperfusion in Septic Patients Undergoing Emergent Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pavlovic Gordana, MD, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NAC11-054(CC11-146)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Abdominal Sepsis; Peritonitis; Colon Perforation
Keywords: Hemoperfusion; Polymyxin-B; Emergency abdominal surgery; Sepsis; Endotoxin
MeSH Terms: conditions — Intraabdominal Infections; Peritonitis; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polymyxin-B hemoperfusion (Active Comparator): In the HEMOPERFUSION group, a veno-venous dialysis catheter type GamCath 12 F, 3 lumen will be inserted instead of a regular double or triple-lumen central venous catheter, and connected to the Toraymyxin® (PMX-20-R) device for endotoxin adsorption by hemoperfusion with the DECAPSMART pump. The length of the hemoperfusion will be a minimum of 120 min and started just before the beginning of the surgical intervention in the OR and stopped at the end of surgery.
  Interventions: Other: Polymyxin-B hemoperfusion
- Control (Active Comparator): In the CONTROL group, the administration of fluids (250 to 500ml crystalloids) and cardiovascular supportive drugs will be guided to maintain standard pressure-related parameters within a normal range: MAP > 65mmHg, HR < 90/min, CVP between > 8 and 12 < mmHg, urinary output > 0.5 ml/kg/h. In line with the conventional approach, other physiological parameters will also be targeted: T° > 35.5°C, Sp02 > 95%, lactate < 2.5 mMol/L, normalisation of the BE.
  At the discretion of the attending anaesthesiologist with the FMH level, a PiCCO monitoring, a transoesophageal echography, or a pulmonary artery catheter, will be inserted to complement the standard hemodynamic monitoring if deemed necessary.
  Interventions: Other: Control

INTERVENTIONS:
Other: Polymyxin-B hemoperfusion
  Arms: Polymyxin-B hemoperfusion
Other: Control
  Arms: Control

SUMMARY:
Septic shock of intra-abdominal origin is likely due to Gram-negative bacteria or mixed pathogens and associated with high levels of endotoxin. The injury to the endothelium results in an increase of endothelial permeability, interstitial edema and release of nitric oxide (NO) that is a very potent vasodilatator. [6] Polymyxins obtained from the Gram-positive bacterium Bacillus polymyxa are antibiotics known for their ability to bind LPS in the outer membrane of the Gram-negative bacterial cell wall as well as free endotoxins with high affinity. Polymyxin-B has been shown to block the activation of cells by a wide variety of LPS. Studies converged to show an improvement in the treatment of septic shock by removing circulating endotoxin.Starting Polymyxin-B hemoperfusion during the operative time is to block the initiation of various deleterious biological cascades induced by endotoxemia such as systemic inflammation, disseminated coagulation disorders, and shock, leading to organ dysfunction and death.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Severe sepsis*or septic shock as define by the ACCCP/SCCM consensus conference, of abdominal origin
* Need for emergent abdominal surgery procedure under general anesthesia with expected duration of ≥ 120 min (in and out patients) for bowel perforation, ileus or peritonitis

Exclusion Criteria:

* Patients younger than 18 years
* Organ transplantation in the last year
* Terminally ill patients: do-not-resuscitate order, perceived to die within 48 hrs of admission
* Known pregnancy or diagnosed by US or Ct-scan (>14 weeks)
* History of sensitivity to polymyxin-B or to anticoagulant ( heparin)
* Uncontrolled hemorrhage within the last 24h
* Severe granulocytopenia ( leukocyte count of < 500/µL)
* Severe thrombocytopenia ( platelets count of < 30'000/µL)
* Need for CPR pre-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be requirement of vasopressors during the first 72 hrs after the beginning of the PMX hemoperfusion using the "inotropic score" | The inotropic score is assessed at the following specific time points: Time 0 - baseline measurements at the beginning of surgery, second time point at the end of surgery, Time 0 +6 hours, Time 0 + 24 hours, Time 0 + 48 hours, Time 0 + 72 hours.

SECONDARY OUTCOMES:
The secondary endpoint will be the variation of MAP, during the first 72 hrs after the beginning of the PMX hemoperfusion | The inotropic score is assessed at the following specific time points: Time 0 - baseline measurements at the beginning of surgery, second time point at the end of surgery, Time 0 +6 hours, Time 0 + 24 hours, Time 0 + 48 hours, Time 0 + 72 hours.
The secondary endpoint will be the variation of "vasopressor dependency index", during the first 72 hrs after the beginning of the PMX hemoperfusion | The variation of the "vasopressor dependency index" is assessed at: Time 0 - baseline measurements at the beginning of surgery, second time point at the end of surgery, Time 0 +6 hours, Time 0 + 24 hours, Time 0 + 48 hours, Time 0 + 72 hours.
The secondary endpoint will be the variation of Pa02/Fi02, during the first 72 hrs after the beginning of the PMX hemoperfusion | The variation of Pa02/Fi02 is assessed at the following specific time points: Time 0 - baseline measurements at the beginning of surgery, second time point at the end of surgery, Time 0 +6 hours, Time 0 + 24 hours, Time 0 + 48 hours, Time 0 + 72 hours.
The secondary endpoint will be the variations of the total SOFA score during the first 7 days after the beginning of the PMX hemoperfusion | The variations of the total SOFA score will be assessed once a day from day 1, till discharge of the ICU, and this maximaly 7 days after the beginning of the PMX hemoperfusion
The secondary endpoint will be the 28-days mortality | The 28-days mortality will be assessed on the 28th day post PMX hemoperfusion
The secondary endpoint will be the 90-days mortality | The 90-days mortality will be assessed on day 90 post PMX hemoperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Pugin, Professor, Study Director — University Hospital, Geneva
Locations (1):
- Emergency operating room, Geneva Cantonal Hospital, Geneva, Switzerland